CLINICAL TRIAL: NCT02938897
Title: A Pilot Randomized Controlled Trial of a Home Telenutrition Weight Loss Program in Men
Brief Title: Telenutrition Weight Loss Study for Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Melissa Ventura-Marra, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1501549080
Record Dates: First submitted 2016-09-25; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Weight Loss; Men
Keywords: Telehealth; Weight loss; Diet quality; Behavioral counseling
MeSH Terms: conditions — Obesity; Weight Loss; Multiple Endocrine Neoplasia Type 1 | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telenutrition Intervention (Experimental): Participants receive diet-related educational materials and self-monitoring tools PLUS registered dietitian nutritionist support.
  Interventions: Behavioral: Registered Dietitian Nutritionist (RDN) Support; Behavioral: Diet-related educational materials; Behavioral: Self-monitoring tools
- Enhanced Usual Care Control (Active Comparator): Participants receive diet-related educational materials and self-monitoring tools.
  Interventions: Behavioral: Diet-related educational materials; Behavioral: Self-monitoring tools

INTERVENTIONS:
Behavioral: Registered Dietitian Nutritionist (RDN) Support — RDN provided individualized medical nutrition therapy via videoconference at weeks 1, 5, and 9 and telephonic nutrition coaching support at weeks 2-4, 6-8, and 10-12.
  Arms: Telenutrition Intervention
Behavioral: Diet-related educational materials — Individualized caloric recommendations (500-750 kcal reduction) were made and food-based educational materials emphasizing general healthful eating patterns and increased intakes of nutrient-rich foods were provided.
Behavioral: Self-monitoring tools — Self-monitoring tools including: weekly weight log, fruit and vegetable tracker, and a SMART (specific, measurable, achievable, relevant, and time bound) goal planner were provided.

SUMMARY:
This study is a 12-week pilot randomized controlled trial to test the feasibility and effectiveness of a home telenutrition weight loss program in men in West Virginia.

DETAILED DESCRIPTION:
This study is a 12-week pilot randomized controlled trial of a home telenutrition weight loss program for men with obesity and at least one additional risk factor for cardiovascular disease. The primary aims are to:

1. To assess the feasibility and acceptability of the male-targeted telenutrition weight loss program in terms of recruitment, retention and satisfaction and
2. To evaluate the effectiveness of the telenutrition program compared to usual care (informational only) with regard to primary and secondary outcome measures at 12 weeks. We hypothesized that men receiving virtual and telephonic support from a registered dietitian nutritionist would have greater weight loss and greater improvements in diet quality than men who were only provided educational materials.

ELIGIBILITY:
Inclusion Criteria:

* 40-70 year old man
* Body mass index ≥ 30
* Living with spouse or companion
* At least one of the following: hypertension, diabetes, pre-diabetes, hypercholesterolemia or hypertriglyceridemia
* A home computer with high-speed internet access
* A telephone for health coach phone calls

Exclusion Criteria:

* Cancer (except skin or prostate), celiac disease, bacterial or viral infections, renal or liver disease (except non-alcoholic fatty liver disease), or condition that prevents fruits and vegetable consumption
* Major surgery or health event (e.g., stroke, heart attack) in the past six months
* Taking insulin, anti-obesity medications, steroids (e.g., Prednisone), or warfarin (Coumadin)
* Pacemaker or defibrillator
* Currently on a weight loss diet or lost > 10 pounds in past six months
* Consume more than two alcoholic beverages daily

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline to 12 weeks

SECONDARY OUTCOMES:
Change in Waist Circumference | Baseline to 6 and 12 weeks
Change in Caloric Intake | Baseline to 6 and 12 Weeks
Change in Diet and Diet Quality | Baseline to 6 and 12 Weeks
  4-day food records, Healthy Eating Index-2010.
Change in Body Composition | Baseline to 6 and 12 Weeks
  Bioelectrical impedance analysis
Health Related Quality of Life | Baseline and 12 Weeks
  HRQOL-4
Program Satisfaction | 6 and 12 Weeks
  Questionnaire
Program Usefulness | 6 and 12 Weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Melissa D Ventura-Marra, PhD, Principal Investigator — West Virginia University

IPD SHARING:
Plan to Share IPD: No
Data will only be reported in aggregate.